CLINICAL TRIAL: NCT06556693
Title: Janus II: A Feasibility Study to Evaluate Response to Remede Dual Channel System Therapy
Brief Title: Janus II Feasibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP3429
Record Dates: First submitted 2024-08-08; First posted 2024-08-16 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention group (Experimental)
  Interventions: Device: Dual Channel Stimulation

INTERVENTIONS:
Device: Dual Channel Stimulation — implant of dual channel stimulation device

SUMMARY:
The objectives of this study are to evaluate the feasibility of the remedē® Dual Channel System at implant and overnight sleep studies and to assess chronic safety.

ELIGIBILITY:
Inclusion Criteria:

* Severe sleep disordered breathing
* Expected to tolerate study procedures
* No heart failure or medically stable heart failure

Exclusion Criteria:

* Currently implanted with a neurostimulator to treat sleep disordered breathing without sponsor approval
* History of severe COPD or pulmonary arterial hypertension
* Current or previous history of nerve injury or palsy
* Prior cervical surgeries or radiation treatment to head region
* Known need for an MRI
* History of psychosis or severe bipolar disorder
* Active Infection or sepsis within 30 days of enrollment
* Currently on kidney dialysis or significantly reduced kidney function
* Hemoglobin less than 8g/dl
* Pacemaker dependance
* New defibrillator or any implantable device or device generator changeout within 30 days prior to study implant or anticipated within the first 12 months
* Other conditions or anticipated surgical procedure expected to affect ability to complete study procedures
* Allergy to contrast dye unless can be prophylactically treated
* Known pregnancy or planning to become pregnant

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Safety through 12 months | 12 Months post implant
  Serious adverse event related to implant procedure, device, or stimulation
Successful Implantation | implant procedure
  Successful Implantation of dual channel system
Improvement in sleep disordered breathing | 12 months post implant
  Demonstration of the acute prevention of sleep disordered breathing events during attended sleep study.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Germany, MD, Study Director — ZOLL Respicardia
Locations (3):
- United States (3):
  - The Insomnia and Sleep Institute of Arizona LLC, Scottsdale, Arizona
  - The University of Michigan Health-West, Wyoming, Michigan
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No